CLINICAL TRIAL: NCT03878927
Title: Phase I Trial, With an Expansion Cohort, of CPX-351 (Cytarabine:Daunorubicin) Liposome Injection in Combination With Gemtuzumab in Subjects With Acute Myeloid Leukemia >55 Years of Age Who Have Not Been Treated With Intensive Chemotherapy
Brief Title: CPX-351+GO in Subjects 55 Years Old, or Older, With AML
Acronym: CPX GO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dose limiting toxicities.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Jazz Pharmaceuticals (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1801018937
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2021-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; De novo AML; Secondary AML; Therapy-related AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): CPX-351 : Daunorubicin 44mg/m^2 and cytarabine 100mg/m^2/day on Days 1,3 and 5 (90 minute IV infusion)
  Gemtuzumab ozogamicin: 3mg/m^2/day on Day 1 (2 hour IV infusion)
  Interventions: Drug: CPX-351; Drug: Gemtuzumab Ozogamicin
- Cohort B (Experimental): CPX-351: Daunorubicin 44mg/m^2 and cytarabine 100mg/m^2 on Days 1, 3 and 5 (90 minute IV infusion)
  Gemtuzumab ozogamicin: 3mg/m^2 on Days 1, 4 (2 hour IV infusion)
  Interventions: Drug: CPX-351
- Cohort C (Experimental): CPX-351: Daunorubicin 44mg/m^2 and cytarabine 100mg/m^2 on Days 1, 3, and 5 (90 minute IV infusion)
  Gemtuzumab ozogamicin: 3mg/m^2 on Days 1, 4 and 7 (2 hour IV infusion)
  Interventions: Drug: CPX-351; Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: CPX-351 — CPX-351 is a liposomal formulation of a fixed combination of the antineoplastic drugs cytarabine and daunorubicin. The two drugs are present inside the liposome in a 5:1 molar ratio. The liposome membrane is composed of distearoylphosphatidylcholine, distearoylphosphatidylglycerol and cholesterol in a 7:2:1 molar ratio.
  Other Names: Vyxeos
Drug: Gemtuzumab Ozogamicin — Gemtuzumab ozogamicin is a CD-33 directed antibody drug conjugated to calicheamicin. CD 33 is expressed on myeloid leukemic blast cells and on normal hematopoietic cells. The drug is approved for the treatment of newly diagnosed CD 33 positive AML in adults and the treatment of relapsed and refractory CD 33 positive AML in adults. The drug is available for injection 4.5 mg as a lyophilized cake or powder in a single use vial for reconstitution and dilution.
  Other Names: Mylotarg
  Arms: Cohort A; Cohort C

SUMMARY:
This is an open label study to assess the safety and efficacy of CPX-351 in combination with gemtuzumab ozogamicin (GO) as first intensive therapy in older (age >55 years) subjects with newly diagnosed AML who are eligible for intensive induction chemotherapy, or AML subjects who previously failed low-intensity therapy but who would be eligible for high-intensity chemotherapy, with companion cognitive function testing to determine whether this contributes to outcome in these subjects. Subjects may have received prior AML treatment with non-intensive regimens, e.g. hypomethylating agents, low-dose cytarabine, or lenalidomide or a clinical trial drug in combination with hypomethylating agents or low-dose cytarabine, but may not have received intensive AML treatment with anthracyclines and/or infusional cytarabine prior to enrollment on this trial. Subjects may not have been treated with GO or other antibody targeting CD 33 prior to enrollment on this trial. The cohort will include 30 subjects treated with the combination of CPX-351 and GO and is designed to establish the safety and feasibility of the combination. These subjects will be assessed for efficacy and safety. Quality of life will be assessed using the FACT-LEU in all subjects. Cognitive function will be assessed using the Blessed Orientation-Memory-Concentration Test and the Montreal Cognitive Assessment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily give informed consent
* Age≥55 years at the time of study treatment
* Pathological diagnosis of AML according to WHO criteria (with >20% blasts in the peripheral blood or bone marrow) including:

  * De novo AML with intermediate or adverse-risk karyotypes (including subjects with karyotypic abnormalities characteristic of MDS), who may have received treatment with low-dose cytarabine, hypomethylating agents, and/or non-intensive chemotherapy-based clinical trial treatments
  * Secondary AML: transformed from prior MDS or MPN, confirmed by bone marrow documentation of prior antecedent hematologic disorder
  * Therapy-related AML: t-AML, requires documented history of prior cytotoxic therapy or ionizing radiotherapy for an unrelated disease
  * Performance status >50% KPS, ECOG 0-2
* Laboratory values fulfilling the following:

  * Peripheral blast count is less than 30,000/μL prior to administration of drug
  * Serum creatinine < 2.5 mg/dL
  * Serum total bilirubin < 2.5 mg/dL
  * Serum alanine aminotransferase or aspartate aminotransferase < 3 times the ULN
  * Subjects with elevated liver enzymes and serum creatinine values secondary to AML are eligible after discussion with PI
  * Cardiac ejection fraction ≥ 50% by echocardiography, MUGA, or Cardiac MRI
  * Negative pregnancy test for non-menopausal women ≥ 55 years old
* Subjects with history of second malignancies in remission may be eligible if there is clinical evidence of disease stability off cytotoxic chemotherapy, documented by imaging, tumor marker studies, etc., at screening. Subjects maintained on long-term non-chemotherapy treatment, e.g., hormonal therapy, are eligible.

Exclusion Criteria:

* Acute promyelocytic leukemia [t(15;17)], AML with karyotype inversion 16 or t(8;21)
* Clinical or morphologic evidence of active CNS leukemia
* Prior intensive chemotherapy for AML with anthracycline/cytarabine-based regimens, GO or other antibody targeting CD33 as a single agent and/ or prior HSCT. Subjects may have been treated with commercially available or investigational hypomethylating agents (e.g. decitabine, azacitidine, SGI-110), lenalidomide, or low-dose cytarabine (not to exceed 20 mg/m2 daily for 14 days for ≤ 6 cycles) or on clinical trials with combinations of low-intensity chemotherapy agents. No more than one agent or combination of agents can be given for treatment of AML prior to enrollment onto this protocol.
* Prior treatment including HMA, systemic chemotherapy, surgery, or radiation therapy must have been completed at least 7 days before start of study treatment or after discussion with PI. Treatment with investigational agents must have been completed at least 14 days prior to study drug treatment. Hydroxyurea is permitted for control of blood counts before the start of study treatment. Toxicities associated with prior therapies must have recovered to grade 1 or less prior to start of study treatment.
* Subjects with prior cumulative anthracycline exposure of greater than 368 mg/m2 daunorubicin (or equivalent).
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent obtaining informed consent
* Subjects with myocardial impairment of any cause (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV staging)
* Active or uncontrolled infection. Subjects with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for ≥72 hrs.
* Subjects with current or recent evidence of invasive fungal infection (blood or tissue culture); subjects with recent fungal infection must have a subsequent negative cultures to be eligible
* Known HIV (new testing not required) or evidence of active hepatitis B or C infection (with rising transaminase values)
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-metabolism disorder
* History of prior bone marrow or solid organ transplantation

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Feasible dose of Gemtuzumab Ozogamicin (GO) in combination with CPX-351 (cytarabine:daunorubicin) in older subjects with AML | 5 years
  The combination of CPX-351 + GO will be declared feasible if at least one dose of GO (day 1, 4, and 7) at 3 mg/m^2 can be safely delivered to subjects.

SECONDARY OUTCOMES:
Efficacy of the combination of CPX and GO as first intensive therapy in elderly (age ≥55 years) by response rate | 5 years
  The efficacy of the combination of CPX-351 and GO in this population will be assessed by treatment response rate, as determined by bone marrow analysis at Day 14 of each induction and consolidation, and as needed thereafter, up to 5 years.
Safety of the combination of CPX and GO in elderly (age ≥55 years) subjects with AML by evaluation of the frequency and severity of adverse events. | 5 years
  The safety of CPX-351 in this population will be assessed by evaluation of the frequency and severity of adverse events.
Assessment of Minimal Residual Disease (MRD) response in subjects treated with this combination using multiparameter flow cytometry and next generation sequencing. | 5 years
  MRD is defined as posttherapy persistence of leukemia cells at levels below morphologic detection, and is a prognostic marker of increased risk of relapse and shorter survival in this subject population.
Quality of Life Assessment using the Functional Assessment of Cancer Therapy-Leukemia (FACT-LEU). | 5 years
  Leukemia Subscale (LeuS): Range:0-68. To derive: Subtract the answers from "4" for each of the 17 questions, except #s 11 and 12 (these are added without modification). Add values, multiply by 17 and divide by # of questions answered. FACT-Leu total =PWB+SWB+EWB+FWB+LeuS. Range: 0-176.
Assessment of the relationship of cognitive function to outcome using the Blessed Orientation-Memory-Concentration Test | 5 years
  The relationship of cognitive function to outcome will be assessed using the Blessed Orientation-Memory-Concentration Test. The score for 6 items are multiplied to yield a "weighted" score. The higher the total weighted score, the more likely the patient has cognitive disability. Weight scores totaling greater than 10 are generally accepted as an indication of the presence of clinically meaningful cognitive impairment.
Assessment of the relationship of cognitive function to outcome using the Montreal Cognitive Assessment (MoCA). | 5 years
  The relationship of cognitive function to outcome will be assessed using the MoCA. The MoCA was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points; a score of 26 or above is considered normal.
CPX-351 as a post-remission (consolidation) therapy | 5 years
  The safety of CPX-351 as a post-remission (consolidation) therapy will be assessed by evaluation of the frequency and severity of adverse events.
Rate of morphologic leukemia-free state (MLFS) | 5 years
  The rate of morphologic leukemia-free state (MLFS) will be determined to supplement the efficacy assessment of CPX-351.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen K Ritchie, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dohner H, Estey EH, Amadori S, Appelbaum FR, Buchner T, Burnett AK, Dombret H, Fenaux P, Grimwade D, Larson RA, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz MA, Sierra J, Tallman MS, Lowenberg B, Bloomfield CD; European LeukemiaNet. Diagnosis and management of acute myeloid leukemia in adults: recommendations from an international expert panel, on behalf of the European LeukemiaNet. Blood. 2010 Jan 21;115(3):453-74. doi: 10.1182/blood-2009-07-235358. Epub 2009 Oct 30. PMID 19880497
- [Background] Stone RM, O'Donnell MR, Sekeres MA. Acute myeloid leukemia. Hematology Am Soc Hematol Educ Program. 2004:98-117. doi: 10.1182/asheducation-2004.1.98. PMID 15561679
- [Background] Appelbaum FR, Gundacker H, Head DR, Slovak ML, Willman CL, Godwin JE, Anderson JE, Petersdorf SH. Age and acute myeloid leukemia. Blood. 2006 May 1;107(9):3481-5. doi: 10.1182/blood-2005-09-3724. Epub 2006 Feb 2. PMID 16455952
- [Background] Kantarjian H, O'brien S, Cortes J, Giles F, Faderl S, Jabbour E, Garcia-Manero G, Wierda W, Pierce S, Shan J, Estey E. Results of intensive chemotherapy in 998 patients age 65 years or older with acute myeloid leukemia or high-risk myelodysplastic syndrome: predictive prognostic models for outcome. Cancer. 2006 Mar 1;106(5):1090-8. doi: 10.1002/cncr.21723. PMID 16435386
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054